CLINICAL TRIAL: NCT01255293
Title: A Prospective, Randomized Study Comparing 1000 Centistoke and 5000 Centistoke Silicone Oil Tamponade for Repair of Proliferative Vitreoretinopathy Retinal Detachments and Diabetic Tractional Retinal Detachments
Brief Title: Comparative Study of 1000 Centistoke Versus 5000 Centistoke Silicone Oil for Repair of Complex Retinal Detachments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Atlantic Retina (Other)
Responsible Party: Jason Hsu, Mid Atlantic Retina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAR-3
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Retinal Detachment; Vitrectomy; Proliferative Vitreoretinopathy; Diabetic Retinopathy
Keywords: Retinal detachment; Proliferative vitreoretinopathy; Diabetic retinopathy; Vitrectomy; Silicone oil
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1000 centistoke silicone oil (Active Comparator)
  Interventions: Procedure: 1000 centistoke silicone oil
- 5000 centistoke silicone oil (Active Comparator)
  Interventions: Procedure: 5000 centistoke silicone oil

INTERVENTIONS:
Procedure: 1000 centistoke silicone oil — Patients who are enrolled in the study and have been identified to have a complex retinal detachment requiring silicone oil tamponade may be randomly assigned to receive 1000 centistoke silicone oil.
  Arms: 1000 centistoke silicone oil
Procedure: 5000 centistoke silicone oil — Patients who are enrolled in the study and have been identified to have a complex retinal detachment requiring silicone oil tamponade may be randomly assigned to receive 5000 centistoke silicone oil
  Arms: 5000 centistoke silicone oil

SUMMARY:
The purpose of this study is to assess the retinal redetachment rates with 1000 centistoke versus 5000 centistoke silicone oil tamponade for repair of complex retinal detachments.

DETAILED DESCRIPTION:
As part of retinal detachment surgery, the eye is typically filled with a gas bubble or silicone oil bubble. This bubble acts like a balloon inside the eye and helps to keep the retina pushed back against the eye wall so it can heal in its proper place. Gas bubbles spontaneously dissolve over a few weeks whereas silicone oil remains in the eye until removed with another surgery. When retinal detachments are associated with significant scar tissue on the retinal surface, silicone oil is often used since it can remain filling the eyeball for as long as necessary to help the retina to heal properly in place. Currently, two different types of silicone oil (1000 centistoke and 5000 centistoke) are commercially available and have been approved for use in the eye by the Food and Drug Administration. The goal of the study is to compare the outcomes using these two different types of silicone oil.

The retinal detachment will be repaired in a standard fashion. There will be no difference between the way retinal detachments are repaired in this study compared to those not in this study. Patients will be randomly assigned (like a flip of a coin) to receive one of the types of silicone oil. Both types of oil have very similar characteristics. The primary difference is that one type is thicker (more viscous) than the other, analogous to honey in comparison with maple syrup.

ELIGIBILITY:
Inclusion Criteria:

* Presence of rhegmatogenous retinal detachment or tractional retinal detachment due to grade C or worse proliferative vitreoretinopathy or proliferative diabetic retinopathy.
* Judgment by the investigator that silicone oil tamponade is surgically indicated for appropriate repair of the complex retinal detachment.
* Visual acuity of light perception or better.
* Ability to provide written informed consent and comply with study assessments for the full duration of the study.

Exclusion Criteria:

* Inability to re-attach the retina at the time of surgery.
* Prior trabeculectomy or tube shunt surgery.
* Corneal opacity which limits visualization of the trabecular meshwork.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Retinal redetachment rate | Six months

SECONDARY OUTCOMES:
Best-corrected visual acuity | 6 and 12 months
Silicone oil emulsification rate | Monthly
  Gonioscopy examination will be used at monthly postoperative visits to assess silicone oil emulsification in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387